CLINICAL TRIAL: NCT01303341
Title: A Phase I Trial of Riluzole and Sorafenib in Patients With Advanced Solid Tumors and Melanoma
Brief Title: Riluzole and Sorafenib Tosylate in Treating Patients With Advanced Solid Tumors or Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02597; NCI-2011-02597 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000695355; 090906; 8850 (Other: Rutgers Cancer Institute of New Jersey); 8850 (Other: CTEP); P30CA072720 (NIH); R01CA149627 (NIH); U01CA132194 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Recurrent Melanoma; Refractory Malignant Solid Neoplasm; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — Riluzole; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (riluzole and sorafenib tosylate) (Experimental): Patients receive riluzole PO BID and sorafenib tosylate PO QD or BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Riluzole; Drug: Sorafenib Tosylate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Riluzole — Given PO
  Other Names: Rilutek
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54 9085; BAY 54-9085; BAY 549085; BAY-54-9085; BAY549085; Nexavar; sorafenib

SUMMARY:
This phase I trial studies the side effects and best dose of sorafenib tosylate when given together with riluzole in treating patients with solid tumors or melanoma that has spread to other places in the body and usually cannot be cured or controlled with treatment. Riluzole may stop or slow the growth of tumor cells. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving riluzole together with sorafenib tosylate may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define a safe dose of sorafenib (sorafenib tosylate) to combine with riluzole in the treatment of patients with all types of solid tumors refractory to standard therapy or for whom no standard therapy exists.

SECONDARY OBJECTIVES:

I. To examine the correlation of clinical or radiologic response with signaling through the mitogen-activated protein kinase (MAPK) and phosphoinositide 3-kinase (PI3K)/protein kinase B (AKT) pathways.

II. To determine if response to therapy with riluzole and sorafenib correlates with expression levels of B-cell lymphoma (BCL)-2, myeloid cell leukemia (MCL)-1, or BCL2-like 11 (apoptosis facilitator) (BIM).

III. To characterize the pharmacokinetics of the combination of riluzole with sorafenib and determine if any drug-drug interactions exist.

IV. To evaluate the microvesicle (an inter-cellular communication approach which may cargo proteins, ribonucleic acids [RNAs] and deoxyribonucleic acids [DNAs] to its host cell) quantification difference between pre-treatment and post-treatment peripheral blood samples of patients.

OUTLINE: This is a dose-escalation study of sorafenib tosylate.

Patients receive riluzole orally (PO) twice daily (BID) and sorafenib tosylate PO once daily (QD) or BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up for approximately 2-3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven solid tumors (Phase I) with biopsiable tumor (expansion cohort) refractory to standard therapy or for whom no standard therapy exists or who decline standard therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must be willing and able to sign informed consent
* Unlimited prior therapies are permitted for patients enrolled in the dose escalation phase of the study; patients in the expansion cohort of the study may not have any prior therapy with riluzole or sorafenib and must have biopsiable tumor
* Patients may have measurable or evaluable disease
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* International normalized ratio (INR) =< 1.5 x institutional ULN
* Creatinine =< 2 x ULN
* Patients with brain lesions that have been treated with whole brain radiotherapy and are clinically stable for at least 4 weeks, are not taking steroids and are not receiving enzyme-inducing anticonvulsants will be eligible

Exclusion Criteria:

* Serious concomitant systemic disorders (including active infections) that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* For patients who have received gamma knife or stereotactic radiosurgery, a 2 week washout is required; patients who have had other types of radiotherapy, chemotherapy or biologic agents within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier to =< grade 1; at least 4 weeks must have elapsed since any major surgery; patients with prostate cancer may continue to receive hormonal therapy
* History of allergic reactions attributed to riluzole or sorafenib
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal, barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 2 weeks after discontinuation of riluzole and/or sorafenib; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; pregnant (positive pregnancy test) or lactating patients cannot participate
* Known human immunodeficiency virus (HIV) infection or known history of active hepatitis B or C infection
* Current, recent (within 4 weeks of the first treatment of this study), or planned participation in an experimental drug study (prevention trials are permitted if the trial is not testing a novel experimental agent)
* Cardiac disease: congestive heart failure > class II New York Heart Association (NYHA); patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* History of stroke within six months
* Clinically significant peripheral vascular disease
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Uncontrolled hypertension, defined as systolic blood pressure > 150 mm Hg or diastolic blood pressure > 90 mm Hg, despite optimal medical management
* Active clinically serious infection > Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Any of the following within 6 months prior to first dose of treatment: myocardial infarction, symptomatic coronary artery disease (severe or unstable angina), artery bypass graft, uncontrolled arrhythmias, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolus
* Pulmonary hemorrhage/bleeding event >= CTCAE grade 2 within 4 weeks of first-dose of study drug
* Any other hemorrhage/bleeding event >= CTCAE grade 3 within 4 weeks of first dose of study drug
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery or significant traumatic injury within 4 weeks of first study drug
* The eligibility of patients taking medications that are potent modulators of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4), cytochrome P450, family 2, subfamily B, polypeptide 6 (CYP2B6), subfamily 2, polypeptide 8 (2C8) will be determined following a review of their case by the principal investigator; every effort should be made to switch patients taking such agents or substances to other medications
* Any condition that impairs the patient's ability to swallow whole pills
* Any malabsorption problem
* Anticipation of need for major surgical procedure during the course of the study
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to day 1 of treatment
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures
* Anticoagulation with Lovenox (enoxaparin) is permitted, however, patients on anticoagulation with warfarin are not permitted on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-02-18 (Actual); Primary Completion 2012-05-01 (Actual); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose of sorafenib tosylate and riluzole in patients with all types of solid tumors | 28 days
  Maximum tolerated dose is defined as the first dose level at which exactly 2/6 patients experience dose limiting toxicity, or at which 1/6 experience dose limiting toxicity and (due to de-escalation) at least 2/3 or 3/6 patients treated with the next higher dose level had dose limiting toxicity.

SECONDARY OUTCOMES:
Suppression of MAPK and PI3K/AKT pathways | Up to 3 years
  Will examine the correlation of clinical or radiologic response with signaling.
Change in BCL-2 expression | Baseline to 3 years
  Appropriate parametric (such as paired t-test) or nonparametric (such as Wilcoxon signed rank test) methods will be used.
Change in MCL-1 expression | Baseline to 3 years
  Appropriate parametric (such as paired t-test) or nonparametric (such as Wilcoxon signed rank test) methods will be used.
Change in BIM expression | Baseline to 3 years
  Appropriate parametric (such as paired t-test) or nonparametric (such as Wilcoxon signed rank test) methods will be used.
Pharmacokinetic parameters of the combination of riluzole with sorafenib tosylate | On days 2, 8, 10, and 15 of each course
  Will be assessed from blood samples.
Change in microvesicle quantification | Baseline to 3 years
  Will be assessed from blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Janice M Mehnert, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Spencer KR, Portal DE, Aisner J, Stein MN, Malhotra J, Shih W, Chan N, Silk AW, Ganesan S, Goodin S, Gounder M, Lin H, Li J, Cerchio R, Marinaro C, Chen S, Mehnert JM. A phase I trial of riluzole and sorafenib in patients with advanced solid tumors: CTEP #8850. Oncotarget. 2023 Apr 10;14:302-315. doi: 10.18632/oncotarget.28403. PMID 37036756